CLINICAL TRIAL: NCT04949685
Title: Evaluation of Clinical and Functional Results After Operative Correction of Lesser Toe Deformities
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201909030RIND
Record Dates: First submitted 2021-06-21; First posted 2021-07-02 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2020-10

CONDITIONS: Plantar Plate Tear; Metatarsalgia; Lesser Metatarsophalangeal Joint Instability; Hammer Toe; Surgery; Plantar Plate Repair
MeSH Terms: conditions — Metatarsalgia; Hammer Toe Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- symptomatic plantar plate rupture: plantar plate repair operation for symptomatic lesser metatarsophalangeal joint instability
  Interventions: Procedure: plantar plate repair

INTERVENTIONS:
Procedure: plantar plate repair — surgical repair via dorsal approach of lesser metatarsophalangeal joint general anesthesia

SUMMARY:
The plantar plate is an important static stabilizer of lesser metatarsophalangeal joints, and disruptions of the plantar plate can lead to significant instability and lesser toe deformities.Our study proposes an inexpensive and versatile method for plantar plate repair

DETAILED DESCRIPTION:
A torn plantar plate is small and difficult to access using regular instruments in a restricted operative field. A unique method for plantar plate repairs was used to repair various configurations of plantar plate tears with standard operative instruments that is available in most operating rooms. A retrospective study was performed on patients who underwent operations for lesser MTPJ instability between September 2015 and December 2019. The outcome analysis included the Lesser Metatarsophalangeal-Interphalangeal Scale from the American Orthopedic Foot and Ankle Society (AOFAS) forefoot score, the Visual Analogue Scale score for pain and satisfaction, and answering the question "Would you recommend this procedure to other patients?"

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lesser metatarsophalangeal joint instability
* Clinical diagnosis of metatarsalgia
* Lesser metatarsophalangeal joint instability clinical grades of II to III, which were determined using the drawer test.

Exclusion Criteria:

* Previous operatve treatment of the affected lesser metatarsophalangeal joint.
* Rheumatioid arthritis.
* Neurologic disorders (e.g., parkinsonism, Charcot's neuroarthropathy…etc.).
* Postoperative follow-ups of less than 12 months

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent operations for lesser metatarsophalangeal joint instability between September 2015 and December 2019.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Lesser Metatarsophalangeal-Interphalangeal Scale from the Americans Orthopedic Foot and Ankle Society (AOFAS) forefoot score (0-100 points) | post-operative >12 months
  One of the most widely used PRO measures for foot and ankle conditions is the American Orthopedic Foot and Ankle Society Score (AOFAS).
  Developed in 1994, the clinician-based AOFAS covers four different regions of the foot: The ankle-hindfoot, midfoot, metatarsophalangeal (MTP)-interphalangeal (IP) for the hallux, and MTP-IP for the lesser toes.
  These four anatomic regions have their own version of the AOFAS survey. Each c is designed to be used independent of the others. However, each measure is comprised of nine questions and cover three categories: Pain (40 points), function (50 points) and alignment (10 points). These are all scored together for a total of 100 points.
Visual Analogue Scale score (VAS) for pain (0-10 points) | pre-opreative and post-operative >12 months
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
  In this study, pre-operative VAS score and post-operative score for pain were obtained for evaluating the clinical outcome. "0" means no pain; "10" means very painful.
Visual Analogue Scale score for satisfaction (0-10 points) | post-operative >12 months
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.
  In this study, pre-operative VAS score and post-operative score for satisfaction were obtained for evaluating the clinical outcome. "0" means unsatisfied ; "10" means very satisfied.

SECONDARY OUTCOMES:
hallux valgus angle (degree) | pre-opreative and post-operative >12 months
  Hallux valgus angle is the angle between the axis of the 1st metatarsal and the axis of the proximal phalanx of the 1st toe. It can only be measured on a radiograph performed whilst weight bearing.
  In this study, pre-operative and post-operative hallux valgus angle were obtained for evaluating the operative outcome.
1-2 intermetatarsal angle (degree) | pre-opreative and post-operative >12 months
  1-2 intermetatarsal angle is the angle between the axis of the 1st metatarsal and the axis of the 2nd metatarsal. It can only be measured on a radiograph performed whilst weight bearing.
  In this study, pre-operative and post-operative hallux valgus angle were obtained for evaluating the operative outcome.
Metatarsophalangeal joint angle( for lesser toes, degree) | pre-opreative and post-operative >12 months
  Metatarsophalangeal joint angle is the angle between the axis of the metatarsal and the axis of the proximal phalanx of the lesser toe. It can only be measured on a radiograph performed whilst weight bearing. positive angle indicates a lateral inclination, and negative angle denotes a varus inclination.
  In this study, pre-operative and post-operative hallux valgus angle were obtained for evaluating the operative outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coughlin MJ. Crossover second toe deformity. Foot Ankle. 1987 Aug;8(1):29-39. doi: 10.1177/107110078700800108. PMID 3623359
- [Result] Weil L Jr, Sung W, Weil LS Sr, Malinoski K. Anatomic plantar plate repair using the Weil metatarsal osteotomy approach. Foot Ankle Spec. 2011 Jun;4(3):145-50. doi: 10.1177/1938640010397342. Epub 2011 Mar 18. PMID 21421939
- [Derived] Chang SM, Huang PJ, Farn CJ, Lin SY, Wang CC, Wang CL, Chen PY. A versatile method for dorsal-approach plantar plate repair using standard operative instruments. BMC Musculoskelet Disord. 2022 Jan 3;23(1):11. doi: 10.1186/s12891-021-04951-w. PMID 34980055